CLINICAL TRIAL: NCT06338930
Title: Remote Monitoring of Patients With an Inflammatory Bowel Disease Under no or Maintenance Therapy
Acronym: ROADMAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ROADMAP
Record Dates: First submitted 2024-02-28; First posted 2024-04-01 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-02

CONDITIONS: Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote monitoring group (Experimental): This group will follow the remote monitoring programme.
  Interventions: Other: Remote monitoring
- Control group (No Intervention): This group will be monitored following the standard of care.

INTERVENTIONS:
Other: Remote monitoring — The intervention group will enroll in the remote monitoring programme. In the standard of care patients visit the outpatient clinic every six months. Patients in the control group will remain in the six-monthly follow-up programma, whereas patients in the intervention group will only visit the outpatient clinic two-yearly. The latter group will be monitored remotely via questionnaires, calprotectin analysis (using CalproSmart) and blood analyses. An IBD nurse will evaluate all incomming data and undertake action if necessary.
  Arms: Remote monitoring group

SUMMARY:
Routine follow-up of patients with inflammatory bowel disease (IBD) under stable doses of maintenance therapy or no IBD-related therapy at all, consists of intensive monitoring with prescheduled outpatient visits every six or twelve months. However, many of these patients do not require additional interventions from the IBD specialist during these visits. In addition, patients in long-term remission, often request a less frequent follow-up in the hospital and in consequence a less frequent absence from school or work. In conclusion, these routinely follow-up visits might put unnecessary burden on both healthcare providers and IBD patients, as well as on healthcare resources.

Until now, no clear standard was set for how to organize a remote monitoring programme that is feasible and safe in a large patient population. Despite the possible added value of remote monitoring for IBD patients on stable or no therapy and who are in remission, they are seldomly the targeted population in clinical trials analysing the effects of remote monitoring in IBD. Secondly, a significant reduction in outpatient clinic visits, is often not actively included in the programme, but more an outcome result. Finally, to compose a safe remote monitoring programme, subjective and objective parameters of disease activity should be collected.

With the ROADMAP study, the main objective is to evaluate the safety and feasibility of remote monitoring in IBD patients that are stable on their current therapy or receive no IBD-related therapy. Secondly, a health economic evaluation will be conducted. Patients will be randomised to either the remote monitoring group or control group. The remote monitoring group will visit the outpatient clinic after two years. During this two-year period, patients will be monitored remotely via three-monthly questionnaires (PRO-2, IBD disk, WPAI, EQ-5D-5L) and faecal calprotectin measures. An IBD nurse will evaluate all incoming data and act in case of red flags.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this Trial must meet all of the following criteria:

1. Patients with Crohn's disease, or ulcerative colitis, or IBD type unclassified
2. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
3. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
4. Patients with access to Mynexuzhealth via smartphone or internet
5. Patients must fluently speak, write, read Dutch.
6. Patients under stable treatment with oral mesalamine, thiopurines, methotrexate, subcutaneous biologicals and/or oral small molecules or under no such therapies at all for at least two years
7. Patients having access to mynexuzhealth (plexus hospitals) or HiX (ZOL)
8. Patients willing to perform a home-based fecal calprotectin measurement every three months through CalproSmart or a similar application, or to go to their general practitioner or a hospital close by to perform a classical ELISA to measure fecal calprotectin every three months*
9. Patients willing to go to their general practitioner or a hospital close by to perform a blood test every year*
10. Patients willing to go to their general practitioner or a hospital close by to perform the required three-monthly blood tests in case of treatment with thiopurines or methotrexate (evaluation of liver tests and complete blood count)*

    * On the day of the classical outpatient clinic organized every two years, this can be performed at UZ Leuven All participants that are considered for Trial participation, per the above criteria will be documented via applicable log forms in Investigator Site File (including Screen Failures).

Exclusion Criteria:

Participants eligible for this Trial must not meet any of the following criteria:

1. Patients receiving an intravenous biological therapy or any form of corticosteroids (with the exception of inhaled or dermatological corticosteroids) in the last two years,
2. Patients with a change in concomitant IBD therapies in the last two years (except for rectal therapies),
3. Patients with IBD-related surgery in the past two years,
4. Patients in whom the IBD team estimates that a more frequent follow-up is required (e.g., due to previous non-compliance, need for additional support, comorbidities such as primary sclerosing cholangitis, cancer, …)
5. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
6. Pregnant patients at screening should be excluded. If the participant becomes pregnant during the study, case-by-case will be evaluated. Study participation or stop should be a mutual decision after clear discussion between physician and patient.

Participants who meet one or more of the above exclusion criteria must not proceed to be enrolled/randomized in the Trial and will be identified via applicable log forms in Investigator Site File.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Patient safety measured as the number of patients not requiring unplanned IBD related hospital visits (outpatient clinic, emergency department, hospitalization, or surgery) or rescue therapy with steroids within two years. | Two years
  Non-inferiority trial: patient safety in the remote monitoring programme must be at least equal to patient safety in standard of care.

SECONDARY OUTCOMES:
Costs and cost savings for hospital, RIZIV, employer, patient, … in the intervention group versus the control group. | Two years
  costs and cost savings
Time saving for patients in the intervention group versus the control group will be measured using a "timing questionnaire". | Two years
  Time savings
Number of telephone/email contacts with the IBD team within one year and within two years. | Two years
  Contact moments with IBD team
Number of contacts with the general practitioner for IBD related reasons within one year and within two years. | Two years
  Number of contacts with GP
Absence at work or school within one year and within two years in the intervention group versus the control group will be measured using the WPAI IBD questionnaire. | Two years
  WPAI
Quality of life in the intervention group versus the control group will be measured using the European Quality of Live Five Dimension Five Level Scale. | Two years
  European Quality of Live Five Dimension Five Level Scale: Aside from general questions regarding the patient's wellbeing, this questionnaire also contains a scale on which "current health" has to be scored with a score between 0 (verry sick) and 100 (perfect health).
Number of patients refusing to participate in this trial and the reason why. | Two years
  Patients refusing to participate and reason
Reasons to stop remote monitoring. | Two years
  The patient can always withdraw consent for participation in the ROADMAP study. In such a case, the investigator will try to collect information on the reason for withdrawing consent.
  Another reason to stop remote monitoring might be that the treating physician decided that it was safer and in the best interest of the patient to stop the remote monitoring programme.
Patient's compliance, measured via missing data in the intervention versus the control group | Two years
  * Number of patients filling out the PRO questionnaire every three months.
  * Number of patients with a fecal calprotectin analysis every three months.
  * Number of patients with a blood test performed every year / three months (in case of patients under thiopurines or methotrexate).
Satisfaction with the program in the intervention group. | Two years
  Patient satisfaction questionnaire. We will ask patients about their satisfaction with the remote monitoring programme.
System usability in the intervention group. | Two years
  System usability scale: is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability. Each question has to be scored with a score of 1 (strongly disagree) to 5 (strongly agree). A high total score, means high system usability.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, Principal Investigator — UZ Leuven

IPD SHARING:
Plan to Share IPD: No